CLINICAL TRIAL: NCT04279613
Title: A Multiple Ascending Dose Trial Investigating Safety, Tolerability and Pharmacokinetics of NNC0361-0041 Administered Subcutaneously to Patients With Type 1 Diabetes Mellitus
Brief Title: A Multiple Ascending Dose Trial Investigating Safety, Tolerability and Pharmacokinetics of NNC0361-0041
Acronym: TOPPLE T1D
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: TN27 Immunoplasmid Therapy; UC4DK117009 (NIH)
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Type I Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: The trial is a placebo-controlled, double-blinded within cohorts, randomized, multiple ascending dose trial with a sequential trial design. A total of 48 patients with T1D are planned to be studied in 4 cohorts of 12 patients (9 on active and 3 on placebo treatment).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NNC0361-0041 (Experimental): Dosage form: 9 mg/ml Solution for injection Route of administration: Subcutaneous Initial dose/Unit dose strength(s)/Dosage level(s) in cohort 1: 1mg Additional doses in cohorts 2, 3, and 4: 5mg, 12.5mg and 25mg Dosing instructions: Once weekly on site
  Interventions: Drug: NNC0361-0041
- Placebo (Placebo Comparator): Dosage form: Solution for injection Route of administration: Subcutaneous Dosing instructions: Once weekly on site
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NNC0361-0041 — Recombinant supercoiled plasmid encoding four human proteins: (pre-proinsulin (PPI), transforming growth factor β1 (TGF-β1), interleukin-10 (IL-10), and interleukin-2 (IL-2) is administered s.c. via syringe and needle.
  Arms: NNC0361-0041
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The trial is a placebo-controlled, double-blinded within cohorts, randomized, multiple ascending dose trial with a sequential trial design. The primary outcome is to investigate the safety and tolerability of ascending subcutaneous weekly doses of NNC0361-0041 plasmid in patients with T1D.

DETAILED DESCRIPTION:
A total of 48 patients with T1D are planned to be studied in 4 cohorts of 12 patients (9 on active and 3 on placebo treatment). Within each cohort, sentinel enrollment will occur and safety assessment will occur before remaining participants are enrolled. The treatment period will be 12 weeks with once weekly dosing leading to 12 doses in total. Dose escalation will occur after data safety review (as described in section 4.9.2). An MMTT to assess insulin secretion will be done at baseline, 1, 3, 6, and 12 months. The follow-up (FU) period will be 1 week after the last dose, as well as 4, 6 and 12 months after the first dose.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide Informed Consent
2. Participants must live in a location with rapid access to emergency medical services
3. Age 18-45 years (both inclusive) at the time of signing informed consent
4. Must have a diagnosis of T1D for less than 48 months at randomization
5. Must have at least one diabetes-related autoantibody present (GAD65A; mIAA, if obtained within 10 days of the onset of insulin therapy; IA-2A; ICA; or ZnT8A)
6. Must have stimulated C-peptide levels greater than or equal to 0.2 pmol/ml measured during an MMTT conducted at least 21 days from diagnosis of diabetes and within one month (37 days) of randomization
7. Be willing to comply with intensive diabetes management
8. HbA1c ≤8.5% at screening
9. Subjects who are CMV and/or EBV seronegative at screening must be CMV and/or EBV PCR negative within 37 days of randomization and may not have had signs or symptoms of a CMV and/or EBV compatible illness lasting longer than 7 days within 37 days of randomization
10. Be up to date on recommended immunizations
11. Be at least 6 weeks from last live immunization
12. Be at least 4 weeks from killed vaccine other than flu vaccine
13. Participants are required to receive killed influenza vaccination at least 2 weeks prior to randomization when vaccine for the current or upcoming flu season is available
14. Be willing and medically acceptable to postpone live vaccines during the treatment period and for 3 months following last dose of study drug
15. If participant is female with reproductive potential, she must have a negative pregnancy test at screening and be willing to avoid pregnancy using a highly effective contraceptive method for the 12 months of the study
16. Males of reproductive age must use adequate contraceptive method during the treatment phase and for 3 months following last dose of study drug
17. Participants are required to receive an authorized non-live COVID-19 vaccination and be fully vaccinated, including eligible boosters as indicated, at least two weeks prior to randomization.

Exclusion Criteria:

Potential participants must not meet any of the following exclusion criteria:

1. One or more screening laboratory values as stated

   1. Leukocytes < 3,000/μL
   2. Neutrophils <1,500 /μL
   3. Lymphocytes <800 /μL
   4. Platelets <100,000 /μL
   5. Haemoglobin <6.2 mmol/L (10.0 g/dL)
   6. Potassium >5.5 mmol/L or <3.0 mmol/L
   7. Sodium >150mmol/L or < 130mmol/L
   8. AST or ALT ≥2.5 times the upper limits of normal
   9. Bilirubin ≥ 1.5 times upper limit of normal
   10. Glomerular Filtration Rate (eGFR) value of eGFR < 60 ml/min/1.73 m2 as defined by KDIGO 2012 (43)
   11. Any other laboratory abnormality that might, in the judgment of the investigator, place the subject at unacceptable risk for participation in this trial
2. Current or ongoing use of non-insulin pharmaceuticals that affect glycemic control within prior 7 days of screening
3. Use of other immunosuppressive agents including chronic use of systemic steroids. Topical products are acceptable (nasal, conjunctival, skin)
4. Have active signs or symptoms of acute infection at the time of randomization
5. Have current, confirmed COVID-19 infection
6. Chronic active infection other than localized skin infections
7. Have evidence of prior or current tuberculosis infection as assessed by PPD, interferon gamma release assay or by history
8. Have evidence of current or past HIV, Hepatitis B infection
9. Have evidence of active Hepatitis C infection
10. Vaccination with a live virus within the last 6 weeks and killed vaccine within 4 weeks (except 2 weeks for flu vaccine)
11. Be currently pregnant or lactating, or anticipate getting pregnant within the one-year study period.
12. Have severe obesity: adults BMI ≥ 40
13. Have a history of malignancies
14. Untreated hypothyroidism or active Graves' disease
15. History of severe reaction to prior vaccination
16. Participation in any clinical trial of an approved or non-approved investigational medicinal product within 30 days after last blood draw (or 5 half-lives of investigational drug, whichever is greater) before screening, or currently enrolled in any other clinical trial
17. Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the trial
18. Supine blood pressure at screening outside the range of 90-139 mmHg for systolic or 50-89 mmHg for diastolic. To exclude white-coat nervousness a single repeat measurement is allowed
19. Have any complicating medical issues or abnormal clinical laboratory results that may interfere with study conduct, or cause increased risk
20. Any condition that in the investigator's opinion may adversely affect study participation or may compromise the study results

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Goland, MD, Study Chair — Type 1 Diabetes TrialNet; Carla Greenbaum, MD, Study Director — Type 1 Diabetes TrialNet
Locations (16):
- United States (16):
  - Children's Hospital of Orange County, Orange, California
  - University of California - San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Barbara Davis Center at University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Indiana University - Riley Hospital for Children, Indianapolis, Indiana
  - Joslin Diabetes Center, Boston, Massachusetts
  - Regents of the University of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - The Naomi Berrie Diabetes Center at Columbia University Medical Center, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Eskind Diabetes Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Benaroya Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data will be available at the National Institute of Diabetes Digestive and Kidney Diseases (NIDDK) Central Repository
URL: https://repository.niddk.nih.gov/home/

REFERENCES:
- [Derived] Pagni PP, Chaplin J, Wijaranakula M, Wesley JD, Granger J, Cracraft J, O'Brien C, Perdue N, Kumar V, Li S, Ratliff SS, Roach A, Misquith A, Chan CL, Coppieters K, von Herrath M. Multicomponent Plasmid Protects Mice From Spontaneous Autoimmune Diabetes. Diabetes. 2021 Aug 13:db210327. doi: 10.2337/db21-0327. Online ahead of print. PMID 34957480
- [Derived] Pagni PP, Chaplin J, Wijaranakula M, Wesley JD, Granger J, Cracraft J, O'Brien C, Perdue N, Kumar V, Li S, Ratliff SS, Roach A, Misquith A, Chan CL, Coppieters K, von Herrath M. Multicomponent Plasmid Protects Mice From Spontaneous Autoimmune Diabetes. Diabetes. 2021 Aug 13;71(1):157-69. doi: 10.2337/db21-0327. Online ahead of print. PMID 34389610

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 mg/0.11 mL NNC0361-0041 Plasmid: Dosage form: 9 mg/ml plasmid in isotonic solution for injection Route of administration: Subcutaneous injection (into the abdomen) Dosing instructions: Once weekly on site for 12 injections Dose/Unit strength in cohort 1: 1mg/0.11 mL
  NNC0361-0041: Recombinant supercoiled plasmid encoding four human proteins: (pre-proinsulin (PPI), transforming growth factor β1 (TGF-β1), interleukin-10 (IL-10), and interleukin-2 (IL-2).
- 5 mg/0.56 mL NNC0361-0041 Plasmid: Dosage form: 9 mg/ml plasmid in isotonic solution for injection Route of administration: Subcutaneous injection (into the abdomen) Dosing instructions: Once weekly on site for 12 injections Dose/Unit strength in cohort 2: 5mg/0.56 mL
  NNC0361-0041: Recombinant supercoiled plasmid encoding four human proteins: (pre-proinsulin (PPI), transforming growth factor β1 (TGF-β1), interleukin-10 (IL-10), and interleukin-2 (IL-2).
- 12.5 mg/1.4 mL NNC0361-0041 Plasmid: Dosage form: 9 mg/ml plasmid in isotonic solution for injection Route of administration: Subcutaneous injection (into the abdomen) Dosing instructions: Once weekly on site for 12 injections Dose/Unit strength in cohort 3: 12.5mg/ 1.4 mL
  NNC0361-0041: Recombinant supercoiled plasmid encoding four human proteins: (pre-proinsulin (PPI), transforming growth factor β1 (TGF-β1), interleukin-10 (IL-10), and interleukin-2 (IL-2).
- 25 mg/2.8 mL NNC0361-0041 Plasmid: Dosage form: 9 mg/ml plasmid in isotonic solution for injection Route of administration: Subcutaneous injection (into the abdomen) Dosing instructions: Once weekly on site for 12 injections Dose/Unit strength in cohort 4: 25mg/2.8 mL
  NNC0361-0041: Recombinant supercoiled plasmid encoding four human proteins: (pre-proinsulin (PPI), transforming growth factor β1 (TGF-β1), interleukin-10 (IL-10), and interleukin-2 (IL-2).
- Placebo: Dosage form: 0 mg/mL Isotonic solution for injection Route of administration: Subcutaneous injection (into the abdomen) Dosing instructions: Once weekly on site for 12 total injections, equivalent volume as prepared IMP
  Placebo: Placebo
Period: Cohort 1: Dose Level 1 mg
Arm/Group | 1 mg/0.11 mL NNC0361-0041 Plasmid | 5 mg/0.56 mL NNC0361-0041 Plasmid | 12.5 mg/1.4 mL NNC0361-0041 Plasmid | 25 mg/2.8 mL NNC0361-0041 Plasmid | Placebo
Started | 9 | 0 | 0 | 0 | 3
Completed | 9 | 0 | 0 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Period: Cohort 2: Dose Level 5 mg
Arm/Group | 1 mg/0.11 mL NNC0361-0041 Plasmid | 5 mg/0.56 mL NNC0361-0041 Plasmid | 12.5 mg/1.4 mL NNC0361-0041 Plasmid | 25 mg/2.8 mL NNC0361-0041 Plasmid | Placebo
Started | 0 | 9 | 0 | 0 | 3
Completed | 0 | 8 | 0 | 0 | 3
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Period: Cohort 3: Dose Level 12.5 mg
Arm/Group | 1 mg/0.11 mL NNC0361-0041 Plasmid | 5 mg/0.56 mL NNC0361-0041 Plasmid | 12.5 mg/1.4 mL NNC0361-0041 Plasmid | 25 mg/2.8 mL NNC0361-0041 Plasmid | Placebo
Started | 0 | 0 | 9 | 0 | 3
Completed | 0 | 0 | 8 | 0 | 3
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Period: Cohort 4: Dose Level 25 mg
Arm/Group | 1 mg/0.11 mL NNC0361-0041 Plasmid | 5 mg/0.56 mL NNC0361-0041 Plasmid | 12.5 mg/1.4 mL NNC0361-0041 Plasmid | 25 mg/2.8 mL NNC0361-0041 Plasmid | Placebo
Started | 0 | 0 | 0 | 8 | 3
Completed | 0 | 0 | 0 | 7 | 2
Not Completed | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 mg/0.11 mL NNC0361-0041 Plasmid | 5 mg/0.56 mL NNC0361-0041 Plasmid | 12.5 mg/1.4 mL NNC0361-0041 Plasmid | 25 mg/2.8 mL NNC0361-0041 Plasmid | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 9 | 8 | 12 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (7.62) | 30.9 (6) | 25.3 (4.57) | 29.5 (7.43) | 29.1 (7.85) | 30.2 (7.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 6 | 4 | 4 | 25
  Male | 3 | 4 | 3 | 4 | 8 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 9 | 9 | 7 | 8 | 12 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 1 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 9 | 6 | 8 | 8 | 11 | 42
  More than one race | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Diagnosis to Randomization [Mean (Standard Deviation); unit: months] | 17.8 (15.3) | 20.2 (12.8) | 10.8 (7.77) | 19 (14.1) | 15.7 (12.6) | 16.6 (12.6)
Weight [Mean (Standard Deviation); unit: kg] | 72.2 (14.4) | 72 (11.5) | 71.9 (11) | 75.9 (13.3) | 79.9 (17.3) | 75.2 (13.5)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.1 (4.43) | 25.6 (3.36) | 24.8 (3.63) | 26 (4.24) | 25.1 (3.73) | 25.1 (3.76)
Autoantibodies positive [Count of Participants; unit: Participants]
  GAD | 9 | 9 | 8 | 7 | 12 | 45
  IA-2 | 2 | 4 | 4 | 7 | 10 | 27
  ICA | 6 | 5 | 4 | 3 | 6 | 24
  Micro-IAA | 5 | 9 | 5 | 7 | 10 | 36
  ZnT8 | 5 | 5 | 4 | 6 | 7 | 27
Count of autoantibodies positive [Count of Participants; unit: Participants]
  1 | 2 | 0 | 1 | 1 | 1 | 5
  2 | 0 | 3 | 2 | 1 | 1 | 7
  3 | 4 | 1 | 4 | 0 | 2 | 11
  4 | 2 | 2 | 2 | 3 | 4 | 13
  5 | 1 | 3 | 0 | 3 | 4 | 11
Glycated hemoglobin level [Mean (Standard Deviation); unit: %] | 6.08 (0.565) | 6.36 (0.922) | 6.01 (0.692) | 6.15 (0.949) | 6.36 (0.817) | 6.21 (0.779)
C-peptide AUC Mean [Mean (Standard Deviation); unit: pmol/mL] | 0.838 (0.385) | 0.645 (0.417) | 0.943 (0.78) | 0.691 (0.623) | 0.753 (0.314) | 0.774 (0.505)
Average total daily dose of Insulin [Mean (Standard Deviation); unit: Units of Insulin] | 22.5 (16.6) | 31.3 (22.5) | 25.8 (14.9) | 26.4 (12.3) | 31.2 (20.7) | 27.9 (17.9)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of adverse events recorded during the on-treatment period, which is defined as from first treatment through visit 15 (or 5 weeks after last treatment for subjects not receiving all injections)
Time Frame: 16 Weeks
Population: The safety analysis set contained all participants who recieved at least one dose of study treatment.
Measure: Number; unit: adverse events
Arm/Group | 1 mg/0.11 mL NNC0361-0041 Plasmid | 5 mg/0.56 mL NNC0361-0041 Plasmid | 12.5 mg/1.4 mL NNC0361-0041 Plasmid | 25 mg/2.8 mL NNC0361-0041 Plasmid | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 8 | 12
adverse events | 230 | 217 | 215 | 169 | 240

2. Secondary Outcome: Change in the Area Under the Plasma C-peptide Concentration-time Curve Across the 2-hour Test Period.
Description: Proportional change from baseline c-peptide AUC mean from a 2-hour mixed meal tolerance test by assessment schedule. The primary outcome is the area under the stimulated C-peptide curve (AUC) based on data collected at time 0 to 2 hours of a 4-hour mixed meal glucose tolerance test (MMTT) conducted at the primary endpoint visit. The timed measurements are done at: 0, 15, 30 60, 90, and 120 minutes. The calculation for the concentration of c-peptide is a weighted average of the 6 timed measurements of c-peptide in nano-moles/Liter. We try to distinguish this calculation from the AUC by referring to it as the "AUC mean" and may be expressed algebraically as the AUC/(120 min.); thus, the units are the same as the y-axis.
Time Frame: 4-, 12-, 24- and 52-weeks from baseline
Population: number of participants analyzed differs in one or more of the rows due to a participant not completing the assessment (MMTT) required to include in computing the geometric mean of the C-peptide change from baseline.
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mL
Arm/Group | 1 mg/0.11 mL NNC0361-0041 Plasmid | 5 mg/0.56 mL NNC0361-0041 Plasmid | 12.5 mg/1.4 mL NNC0361-0041 Plasmid | 25 mg/2.8 mL NNC0361-0041 Plasmid | Placebo
Number analyzed (Participants) | 9 | 8 | 7 | 7 | 10
pmol/mL
  4 weeks | 0.861 [0.741 to 1] | 0.955 [0.729 to 1.25] | 1.15 [0.845 to 1.55] | 0.823 [0.645 to 1.05] | 0.8 [0.695 to 0.921]
  12 weeks | 0.83 [0.724 to 0.95] | 0.807 [0.608 to 1.07] | 0.914 [0.602 to 1.39] | 0.775 [0.646 to 0.931] | 0.794 [0.681 to 0.927]
  24 weeks | 0.761 [0.611 to 0.946] | 0.655 [0.411 to 1.05] | 0.93 [0.704 to 1.23] | 0.809 [0.638 to 1.03] | 0.764 [0.63 to 1]
  52 weeks: number analyzed (Participants) | 8 | 7 | 7 | 7 | 10
  52 weeks | 0.742 [0.549 to 1] | 0.626 [0.467 to 0.841] | 1.01 [0.705 to 1.46] | 0.65 [0.467 to 0.905] | 0.585 [0.495 to 0.692]

ADVERSE EVENTS:
Time Frame: Baseline visit (V0) through week 52 study visit (V17)
Description: From study start through visit 15, all adverse events which were grade 1 or greater per the NCI CTCAE v5.0 were required to be reported. For visits 16 and 17 only grade 2 or greater were to be reported. Hypoglycemia/hyperglycemia only to be reported as AEs in the case of requiring assistance of others due to loss of consciousness/DKA. All SAEs were required to be reported. Adverse events were analyzed based on organ class system without regard to the specific adverse event term.
Arm/Group | 1 mg/0.11 mL NNC0361-0041 Plasmid | 5 mg/0.56 mL NNC0361-0041 Plasmid | 12.5 mg/1.4 mL NNC0361-0041 Plasmid | 25 mg/2.8 mL NNC0361-0041 Plasmid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/8 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 1/9 | 0/8 | 0/12
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9 | 9/9 | 8/8 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg/0.11 mL NNC0361-0041 Plasmid (N=9) | 5 mg/0.56 mL NNC0361-0041 Plasmid (N=9) | 12.5 mg/1.4 mL NNC0361-0041 Plasmid (N=9) | 25 mg/2.8 mL NNC0361-0041 Plasmid (N=8) | Placebo (N=12)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg/0.11 mL NNC0361-0041 Plasmid (N=9) | 5 mg/0.56 mL NNC0361-0041 Plasmid (N=9) | 12.5 mg/1.4 mL NNC0361-0041 Plasmid (N=9) | 25 mg/2.8 mL NNC0361-0041 Plasmid (N=8) | Placebo (N=12)
Investigations (Investigations) | 9 (96) | 9 (143) | 9 (133) | 8 (81) | 12 (134)
Vascular disorders (Vascular disorders) | 8 (46) | 8 (33) | 6 (21) | 7 (21) | 10 (36)
General disorders and administration site conditions (General disorders) | 6 (23) | 2 (9) | 4 (10) | 5 (16) | 7 (19)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 6 (15) | 4 (5) | 3 (5) | 4 (7) | 6 (14)
Infections and infestations (Infections and infestations) | 5 (7) | 5 (6) | 5 (9) | 3 (4) | 3 (3)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (5) | 7 (16) | 6 (10) | 4 (6) | 2 (7)
Gastrointestinal disorders (Gastrointestinal disorders) | 5 (10) | 4 (7) | 3 (9) | 3 (8) | 4 (4)
Nervous system disorders (Nervous system disorders) | 4 (18) | 3 (5) | 3 (10) | 4 (13) | 3 (5)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 5 (13) | 1 (2) | 4 (6) | 2 (3) | 4 (7)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (7) | 2 (3) | 1 (2) | 3 (4) | 5 (5)
Renal and urinary disorders (Renal and urinary disorders) | 6 (8) | 4 (6) | 0 (0) | 1 (3) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (5) | 3 (9) | 4 (7)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 (7) | 2 (2) | 1 (1) | 1 (1) | 3 (4)
Cardiac disorders (Cardiac disorders) | 2 (5) | 1 (1) | 2 (5) | 0 (0) | 3 (5)
Psychiatric disorders (Psychiatric disorders) | 1 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Eye disorders (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Endocrine disorders (Endocrine disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Immune system disorders (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT04279613/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT04279613/SAP_001.pdf